CLINICAL TRIAL: NCT03160365
Title: Innovative Planning and Guidance System for Prostate Focal Brachytherapy
Acronym: FOCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC17.0094 FOCUS
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The patient will have some exams more than in the current way
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACQUISITION OF IMAGES (Other): 4 MRIs were performed at Day 0, day 1, day 15 and day 30 and a preoperative CT scan without injection of a contrast agent.
  Interventions: Procedure: ACQUISITION OF IMAGES

INTERVENTIONS:
Procedure: ACQUISITION OF IMAGES — In addition to the conventional clinical protocol, 4 MRIs qere performed at Day 0, day 1,day 15 and day 30 and a preoperative CT scan without injection of a contrast agent.

SUMMARY:
A key feature of low-dose brachytherapy is that irradiation affects only a local area around the inserted radiation sources. The exposure of healthy tissues around these sources is then reduced. However, the number of adverse events remains high (about 79% of patients with sexual problems and 30% of patients with urinary incontinence) and brachytherapy is no better than other treatment options for Preservation of the urethral apparatus (about 40% of patients).

The current technique for the implantation of radioactive sources, which has not been revised since the early 1980s, consists in imaging the prostate at the beginning of the intraoperative procedure with transrectal ultrasound in order to evaluate the size and shape of the prostate . This information is then used to identify the best distribution of the dose of radiation to be administered to each patient. This treatment planning step is based on a procedure where the operator manually places 50 to 100 grains of iodine in the prostate. These grains are inserted transperinally under transrectal 2D ultrasound control, using needles through a transperineal grid with several needle guides evenly spaced 5 mm apart. This is an arduous task because this manual grain placement procedure must take into account the dose to be administered to the prostate without exceeding the dose limit for the surrounding organs at risk (rectum, urethra). In addition, the overestimation of the dose formality called TG-43 and the inaccurate grain placement can contribute to the creation of cold spots where no dose is administered. It may be responsible for recurrences of prostate cancer after brachytherapy treatment. Although brachytherapy dosimetry has been extensively researched, the TG-43 dose formalism has been the benchmark for the last 20 years. Moreover, from an economic point of view, the high side-effects rates of the treatment of prostate cancer result in particularly expensive post-treatment costs. The search for improved solutions for the treatment of prostate cancer remains a major societal challenge.

In recent years, a very attractive therapeutic alternative between active surveillance and overall treatment is gaining popularity among experts: focal therapy.

It is a localized treatment, limited to cancerous areas, in order to preserve healthy functional tissues inside and outside the organ and thus the quality of life of the patient.

Focal therapy is also often the preferred solution for recovery therapy (second intervention).

Finally, focal therapy has great potential to reduce the cost and duration of the intervention, as well as the cost of follow-up.

In recent years, several energies have been proposed as being adapted to focal therapy, such as high intensity focal ultrasound, laser ablation and cryotherapy. Brachytherapy, which already gives above average results in the treatment of whole glands, has been identified as a very good candidate for this new therapeutic paradigm.

In brachytherapy, radioactive grains are implanted in the prostate using transperineal catheters. The rapid reduction of the dose according to the distance of the radioactive seeds gives the physician a great flexibility to control the radiation accurately. It allows intermediate approaches between global and focal treatments, providing great scalability, and it is a good candidate for recovery therapy.

Recent studies have shown that focal brachytherapy allows more than half of the needles and seeds to act more strongly on the target while irradiating Significantly less The urethra and rectum. Clinical studies on this subject are still limited and further research is needed to confirm the performance of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for prostate brachytherapy
* Male patients, aged at least 18 years with no age limit.
* Prostate adenocarcinoma with proved histology (prostate biopsy)
* Localized disease: Negative extension (TAP + TAP + bone scintigraphy)
* Absence of contraindications to surgery or general anesthesia Prostatic volume less than or equal to 60 cc
* Prognostic group of "low risk" according to the classification of D'Amico (Gleason less than or equal to 6 AND PSA <10ng / ml AND less than or equal to T2a to the rectal touch)
* Prognostic group "favorable intermediate" according to the classification of D'Amico (with no more than one criterion among the following: Gleason 7 (3 + 4), PSA <15ng / ml, less than half of the positive biopsies). Note: Gleason 7 (4 + 3) are excluded.
* Absence of prophylactic capsular collapse on prostatic MRI
* Absence of irritative urinary signs too important
* No history of pelvic irradiation
* Absence of colorectal inflammatory disease in evolutionary thrust
* Informed Consent
* Affiliated to a social security scheme or beneficiary

Exclusion Criteria:

* A protected major person within the meaning of the Public Health Code
* Refus or inability to give informed consent
* NO-indication to CT SCAN and MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Acquisition images | 1 month
  The volume of the prostate was evaluated from acquisition of CT and MRI after brachytherapy which causes an increase of it following the insertion of the needles to create a predictive model.

SECONDARY OUTCOMES:
Adjustement of doses | 1 month
  The dosimetric planning will be adjusted using the predictive model of the evolution of the prostate volume.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No